CLINICAL TRIAL: NCT01234792
Title: Single-Dose Nicotine Pharmacokinetics With Three Oral Nicotine Replacement Products - A Study in Healthy Smokers
Brief Title: Single-dose Nicotine Pharmacokinetics With Three Oral Nicotine Replacement Products. A Study in Healthy Smokers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NICTDP1070; 2008-000596-15 (EudraCT Number)
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Tobacco Dependence
Keywords: Smoking Cessation, Nicotine pharmacokinetics
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Nicotine Chewing Gum

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- NIC-6 (Experimental): 6 mg Experimental nicotine gum
  Interventions: Drug: 6 mg Experimental nicotine gum
- NIC-4 (Active Comparator): 4 mg Nicotine Gum
  Interventions: Drug: 4 mg Nicotine Gum/
- NIC-2 (Active Comparator): 2 mg Nicotine Gum
  Interventions: Drug: 2 mg Nicotine Gum

INTERVENTIONS:
Drug: 6 mg Experimental nicotine gum — A single 6 mg dose of an experimental nicotine gum, with a 36-hour washout between visits
  Other Names: Not marketed
  Arms: NIC-6
Drug: 4 mg Nicotine Gum/ — A single 4 mg dose of Nicorette® gum, with a 36-hour washout between visits
  Other Names: Nicorette® Gum
  Arms: NIC-4
Drug: 2 mg Nicotine Gum — A single 2 mg dose of Nicorette® gum, with a 36-hour washout between visits
  Other Names: Nicorette® Gum
  Arms: NIC-2

SUMMARY:
Single-dose nicotine pharmacokinetics with three oral nicotine replacement products.

DETAILED DESCRIPTION:
The study is a single-dose, randomized, crossover study with 24 subjects (all subjects will receive all treatments). The investigational products will be 6 mg, 4 mg and 2 mg Nicotine medicated gum given as single doses at separate treatment visits. Periods without NRT, lasting for at least 36 hours, will separate treatment visits. Blood for pharmacokinetic analyses will be drawn before, and at 2.5, 5, 7.5, 10, 15, 20, 30, 45, and 60 minutes as well as after 1.5, 2, 4, 6, and 8 hours after start of product administration. Subjects will also be monitored to capture any adverse events that may occur. The trial is blind in the sense that treatment labels will not be revealed to subjects and trial personnel. Also the bioanalysts, pharmacokineticists and monitor will be unaware of treatment labels.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects, smoking at least 15 cigarettes daily during at least one year preceding inclusion and BMI between 17.5 and 30.0 kg/m2 and a total body weight of at least 55.0 kg.
* Female participants of child-bearing potential are required to use a medically acceptable means of birth control.
* A personally signed and dated informed consent document, indicating that the subject has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Pregnancy, lactation or intended pregnancy.
* Treatment with an investigational product or donation or loss of blood within 3 month preceding the first dose of study medication.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | During 8 hours post-dose
  Cmax, which is the maximum observed plasma concentration, measured in nanograms/milliliter (ng/mL)
Area Under the Curve (AUC)(0-t) | During 8 hours post-dose
  AUC(0-t), whitch is the area under the plasma concentration-vs.-time curve from start of drug administration until the time of the last measurable plasma concentration, calculated as hour * nanograms (ng) per milliliter (mL).
AUC(0-∞) | 8 hours post-dose
  AUC(0-∞), which is the area under the plasma concentration-vs.-time curve from start of drug administration until infinity.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kruse, PhD, Study Director — McNeil AB
Locations (1):
- McNeil AB Clinical Pharmacology R&D, Lund, Sweden